CLINICAL TRIAL: NCT03512613
Title: A Pilot Study- Monitoring Cerebral Blood Flow in Neonates With Congenital Heart Defects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ornim Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: RDCL- IL-SMC-021
Record Dates: First submitted 2018-02-22; First posted 2018-05-01 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Congenital Heart Defect; Cerebrovascular Circulation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: c-FLOW 3310-P — c-FLOW 3310-P is a continuous, non-invasive monitor of cerebral deep tissue blood flow used to measure relative changes in blood flow.
  The device monitors regional micro circulatory blood flow in tissues, by using sensors placed near the area of interest.

SUMMARY:
Congenital heart defects have an incidence of 9/1000 live births. Infants with congenital heart defects such as Transposition of Great Arteries / Hypoplastic Left Heart are at risk for brain injury because of concomitant brain malformations. Previous studies of cerebral MRI in infants with congenital heart defects showed that in 20-40% of cases there was preoperative brain injury and post operative with the same incidence. These findings are strongly associated with early and long-term neurodevelopmental injury.

There is a necessity for a non invasive device who will monitor the cerebral blood flow during the hospitalization prior and post the cardiac defect repair surgery.

The previous modal of the study device has been cleared for marketing by the FDA (k150268).

The main goal of this study is to demonstrate that the new design of Ornim's c-FLOW 3310-P is easy to operate and effective in monitoring changes in cerebral blood flow in neonates as demonstrated in adults.

DETAILED DESCRIPTION:
55 eligible neonates whom have been deemed as candidates for a cardiac surgery will be enroll to the study.

At the first phase, 10 neonates will be monitored. After the investigator has assessed the patient as eligible for the study and consent will be received by the parents, the subject will be provided with a study enrollment number.

All clinical assessments routinely preformed as per standard of care during all hospitalization, such as hemodynamic continues parameters, discreet samples will be documented in the medical records, and later on the requested assessments will be recorded in the designated Case Report Form.

Monitoring will be performed a day prior to the repair surgery, following the surgery at the same day and one and two days after, for 3 hours per day.

Additional standard of care parameters will be collected :Heart rate, Mean Arterial Blood Pressure, Saturation, Ventilator rate, Medications, Blood gases ( blood tests), Echocardiogram, pre-surgery Head US,. additional examination will be performed intended for the study: two post surgery Head US, S100B biomarker for brain injury and Neurological examinations prior and 7 days post- surgery( By standardized questionnaires).

Sample size: 55:

A sample size of 55 will enable to detect an increase of 20% in flow with a standard deviation of 50 assuming normal distribution a type 1 error of 5% and power of 80%.

In order to evaluate the study design and data quality the sponsor will perform an interim analysis for the 10 first neonates.

Quality assurance: Following the study initiation monitoring visit will be performed for the first patient. Additional visits will be performed according to recruitment rate. Source data verification and safety events follow up will be performed during those visits.

Plan for missing data: Every effort will be made to complete follow-up for all subjects and avoid missing data, in particular regarding essential items.

Statistical analysis: Descriptive statistics will be used to summarize results. Categorical measurements will be presented in contingency tables with counts & percent.

Continuous measurements will be presented with N, means ±Standard Deviation, or median with 25th & 75th percentiles Minimum & Maximum.

The percent of change in flow pre & post maneuver will be calculated using one sample t-test.

Spearman correlation will be used to correlate the autoregulation index and neurological outcomes.

Significance level will be defined as a=0.05. Statistical analyses will be carried out using SPSS (Statistical Package for the Social Sciences) 24.01 software.

ELIGIBILITY:
Inclusion Criteria:

1. Mutual parents' consent (outstanding exceptional cases who approved by the EC)
2. Born at gestational age of more than 34+6/7 weeks
3. Cardiac surgery between 0- 4 weeks of age
4. Head circumference >= 31 cm

Exclusion Criteria:

1. Patient with implants located in the intended area of the c-FLOW 3310-P sensor location.
2. Laceration of scalp injury at the intended area of the c-FLOW 3310-P sensors
3. Known brain malformation
4. Hydrocephalus
5. Resuscitation between the time of surgery and neurological outcome assessment

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with congenital heart disease scheduled for repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2018-05-29 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in c-Flow3310-P following routine maneuvers | 3 hours monitoring per day, for 4 days
  Changes will be measured following routine maneuvers such as suction, leg lifting, Blood sample, changing position, feeding, presence of feeding tube etc.
  Change= (CFI(manipulation)- CFI(baseline))- CFI(baseline)

SECONDARY OUTCOMES:
The correlation between Auto-regulation index and Neurological outcomes | 3 hours monitoring per day, for 4 days
  Auto regulation index (the correlation of Cerebral Flow Index& Mean Arterial Pressure)
  Neurological outcomes based on two validated questionnaires:
  PCPC (Pediatric Cerebral Performance Category) scale- ranging from 1-6 PSOM ( Pediatric Stroke Outcome Measure) scale - ranging from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bar Yosef, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Govindan RB, Massaro AN, Andescavage NN, Chang T, du Plessis A. Cerebral pressure passivity in newborns with encephalopathy undergoing therapeutic hypothermia. Front Hum Neurosci. 2014 Apr 24;8:266. doi: 10.3389/fnhum.2014.00266. eCollection 2014. PMID 24795612
- [Result] Massaro AN, Govindan RB, Vezina G, Chang T, Andescavage NN, Wang Y, Al-Shargabi T, Metzler M, Harris K, du Plessis AJ. Impaired cerebral autoregulation and brain injury in newborns with hypoxic-ischemic encephalopathy treated with hypothermia. J Neurophysiol. 2015 Aug;114(2):818-24. doi: 10.1152/jn.00353.2015. Epub 2015 Jun 10. PMID 26063779
- [Result] Tsalach A, Ratner E, Lokshin S, Silman Z, Breskin I, Budin N, Kamar M. Cerebral Autoregulation Real-Time Monitoring. PLoS One. 2016 Aug 29;11(8):e0161907. doi: 10.1371/journal.pone.0161907. eCollection 2016. PMID 27571474
- [Result] Hori D, Hogue CW Jr, Shah A, Brown C, Neufeld KJ, Conte JV, Price J, Sciortino C, Max L, Laflam A, Adachi H, Cameron DE, Mandal K. Cerebral Autoregulation Monitoring with Ultrasound-Tagged Near-Infrared Spectroscopy in Cardiac Surgery Patients. Anesth Analg. 2015 Nov;121(5):1187-93. doi: 10.1213/ANE.0000000000000930. PMID 26334746
- [Result] Rachelia, N. (2012). Non-Invasive Blood Flow Measurements Using Ultrasound Modulated Diffused Light. In Photons Plus Ultrasound: Imaging and Sensing 2012.